CLINICAL TRIAL: NCT00586781
Title: Investigational Device Exemption for the Scandinavian Total Ankle Replacement (STAR) - Bilateral Arm
Brief Title: Study of the Scandinavian Total Ankle Replacement (STAR) for the Treatment of Bilateral Degenerative Ankle Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Link America, Inc. (Industry)
Responsible Party: Andrew Greenberg, President, Link America, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Link-3
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-12

CONDITIONS: Osteoarthritis; Post-Traumatic Arthritis; Rheumatoid Arthritis
Keywords: ankle replacement; end-stage arthritis of the ankle; degenerative ankle disease
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3 (Experimental): The S.T.A.R. ankle system is the study device. The device has three parts: two metal bearing surfaces (cobalt-chromium alloy) plates with bars that fit into the bone and one plastic (polyethylene) spacer that moves between the metal plates like a ball bearing. The materials in the S.T.A.R. device are the same materials used in total hip and knee implants. Both ankles of every subject will be treated with the STAR ankle.
  Interventions: Device: Scandinavian Total Ankle Replacement (STAR)

INTERVENTIONS:
Device: Scandinavian Total Ankle Replacement (STAR) — The device has three parts: two metal bearing surfaces (cobalt-chromium alloy) plates with bars that fit into the bone and one plastic (polyethylene) spacer that moves between the metal plates like a ball bearing. The materials in the S.T.A.R. device are the same materials used in total hip and knee implants.

SUMMARY:
The purpose of this study is to evaluate the safety of the S.T.A.R. device for patients with bilateral disease.

DETAILED DESCRIPTION:
The specific objectives are to show that the safety data of the S.T.A.R. ankle arthroplasty is similar for treatment of single ankle disease (as defined in the pivotal study) and bilateral ankle disease. The bilateral disease may be identified at the time of enrollment or may have progressed after enrollment and treatment of the first ankle in the pivotal study.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe pain, loss of mobility and function of the ankle
* Primary arthrosis, post traumatic arthrosis or rheumatoid arthrosis
* At least six months of conservative treatment for severe ankle conditions
* Bilateral ankle disease that have not been enrolled in the pivotal study or single ankle disease and enrolled in the pivotal study but have subsequently developed ankle disease in the contralateral ankle and require surgical intervention
* Willing and able to give informed consent

Exclusion Criteria:

* Patients who have not reached skeletal maturity
* Active or prior deep infection in the ankle joint or adjacent bones
* Prior arthrodesis at the involved site
* History of prior mental illness or patient demonstrates that their mental capacity may interfere with their ability to follow the study protocol
* Obesity (weight greater than 250 lbs)
* History of current or prior drug abuse or alcoholism
* Any physical condition precluding major surgery
* Prior surgery and/or injury that has adversely affected the ankle bone stock
* Severe osteoporotic or osteopenic condition or other conditions that may lead to inadequate implant fixation in the bone
* Insufficient ligament support

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2001-09; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Safety endpoints to be measured are: • Device failure or device removal/revision • Radiographically confirmed loosening and migration • Complications | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roger A Mann, MD, Principal Investigator — Roger A Mann, Inc; Michael J Coughlin, MD, Principal Investigator — Foot and Ankle
Locations (5):
- United States (5):
  - Mayo Clinic, Jacksonville, Florida
  - University of Iowa, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Duke University Medical Center, Durham, North Carolina
  - Orthopedic Associates of Dallas, Dallas, Texas